CLINICAL TRIAL: NCT06883240
Title: A Multicenter Non-Interventional Study Evaluating Bleeds and Health-Related Quality Of Life in Patients With Type 3 Von Willebrand Disease on Prophylactic Standard-of-Care Treatment
Brief Title: An Observational Study of Participants With Type 3 Von Willebrand Disease on Prophylactic Standard-of-Care Treatment
Acronym: WILL-EMI NIS
Status: Recruiting | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: WP45335
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Von Willebrand Disease, Type 3
MeSH Terms: conditions — von Willebrand Disease, Type 3

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants with Type 3 VWD Treated with Prophylactic SOC: Participants with Type 3 VWD, aged 2 years and above, who are currently on standard of care (SOC) prophylactic therapy are anticipated to remain on the chosen SOC regimen during the study. Dosing and treatment duration of any studied medicinal products collected as part of this study are at the discretion of the treating physician in accordance with local labeling or local treatment guidelines.
  Interventions: Drug: Von Willebrand Factor Concentrates; Drug: Von Willebrand Factor Concentrates and Factor VIII Concentrates; Drug: Factor VIII Concentrates; Drug: Recombinant Activated Factor VII; Drug: Activated Prothrombin Complex Concentrate

INTERVENTIONS:
Drug: Von Willebrand Factor Concentrates — Used according to local labeling or local treatment guidelines.
Drug: Von Willebrand Factor Concentrates and Factor VIII Concentrates — Used according to local labeling or local treatment guidelines.
Drug: Factor VIII Concentrates — Used according to local labeling or local treatment guidelines.
Drug: Recombinant Activated Factor VII — Used according to local labeling or local treatment guidelines.
Drug: Activated Prothrombin Complex Concentrate — Used according to local labeling or local treatment guidelines.

SUMMARY:
This non-interventional study (NIS) is designed to collect information on the effectiveness and safety of treatment received in routine clinical care, as well as measure the health-related quality of life (HRQoL) of participants with Type 3 von Willebrand disease (VWD) receiving prophylactic therapy per local standard of care (SOC) over an observation period of at least 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Type 3 von Willebrand disease (VWD), based on medical records
* Adequate hematologic, hepatic, and renal function
* Documented and confirmed previous use of SOC prophylactic therapy for VWD (1-3 times weekly, as per prescribed dose) and anticipation to remain on the same regimen during the study
* For participants of childbearing potential: agreement to remain abstinent or adhere to the contraception requirements

Exclusion Criteria:

* Inherited or acquired bleeding disorder other than Congenital Type 3 VWD
* History of gastrointestinal bleeding within 18 months prior to enrollment, or any previous diagnosis of angiodysplasia
* History of intracranial hemorrhage
* Previous or current treatment for thromboembolic disease or signs of thromboembolic disease
* Other conditions (e.g., certain autoimmune diseases) that may increase risk of bleeding or thrombosis
* History of clinically significant hypersensitivity associated with monoclonal antibody therapies or components of the emicizumab injection
* Use of systemic immunomodulators (e.g., interferon) at enrollment or planned use during the study, with the exception of anti-retroviral therapy

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will observe approximately 40 participants with Type 3 VWD (aged 2 years and older) that are currently being treated with SOC prophylactic therapy.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Annualized Bleed Rate (ABR) for Treated Bleeds | From Baseline to at least 24 weeks

SECONDARY OUTCOMES:
ABR for All Bleeds | From Baseline to at least 24 weeks
ABR for Treated Spontaneous Bleeds | From Baseline to at least 24 weeks
ABR for Treated Joint Bleeds | From Baseline to at least 24 weeks
Incidence and Severity of Adverse Events, with Severity Determined According to the World Health Organization (WHO) Toxicity Grading Scale | From Baseline until study completion (at least 24 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (27):
- United States (4):
  - UC Davis, Sacramento, California
  - University of Florida, Gainesville, Florida
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
- UZ Leuven Gasthuisberg, Leuven, Belgium
- Canada (2):
  - The Hospital for Sick Children, Toronto, Ontario
  - McGill University Health Center, Montreal, Quebec
- IPS SURA Industriales Medellín, Medellín, Colombia
- France (2):
  - Hopital Claude Huriez - CHU Lille, Lille
  - Groupe Hospitalier Necker Enfants Malades, Paris
- Germany (3):
  - Universitätsklinikum Bonn, Bonn
  - Gerinnungszentrum Rhein-Ruhr;Gerinnungsambulanz, Duisburg
  - Hämophiliezentrum Med. Klinik III/Institut für Transfusionsmedizin, Frankfurt/M.
- Italy (3):
  - Universita' Degli Studi La Sapienza-Ist.Di Ematologia, Rome, Lazio
  - IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - AOU Careggi, Florence, Tuscany
- Japan (2):
  - Kurume University Hospital, Fukuoka
  - Tokyo Medical University Hospital, Tokyo
- Erasmus MC, Rotterdam, Netherlands
- Instytut Hematologii i Transfuzjologii, Warsaw, Poland
- Charlotte Maxeke Johannesburg Academic Hospital, Johannesburg, South Africa
- Spain (2):
  - Hospital Universitario la Paz, Madrid
  - Hospital Universtiario Virgen del Rocio, Seville
- Sahlgrenska Universitetssjukhuset, Gothenburg, Sweden
- United Kingdom (3):
  - St Thomas' Hospital, London
  - Great Ormond Street Hospital, London
  - Manchester Royal Infirmary, Manchester

IPD SHARING:
Plan to Share IPD: No